CLINICAL TRIAL: NCT03616093
Title: The Impact of Acute (2 h) and Short-term (4 Days) Nitrate Supplementation in the Form of Red Beet Root Juice on Intense Intermittent Exercise Performance.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PEP-1718
Record Dates: First submitted 2018-06-06; First posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Exercise Performance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Beet shot (Experimental): Active supplement containing 6.2 mmol nitrate
  Interventions: Other: Test Beet Shot
- Placebo beverage (Placebo Comparator): Placebo supplement containing negligible nitrate
  Interventions: Other: Placebo Beverage

INTERVENTIONS:
Other: Test Beet Shot — Active supplement containing 6.2 mmol nitrate
  Arms: Test Beet shot
Other: Placebo Beverage — Placebo supplement containing negligible nitrate
  Arms: Placebo beverage

SUMMARY:
Both acute ingestion (1-3 h) and chronic supplementation (3-30 days) with dietary nitrate has been shown to increase nitric oxide activity and, in some studies, to improve exercise economy, exercise tolerance, and endurance exercise performance. In addition, more recent evidence suggests that dietary nitrate has the potential to enhance team-sport-specific high-intensity intermittent exercise performance. Indeed, chronic dietary nitrate supplementation (2-6 days) has been reported to increase the distance covered before exhaustion during the Yo-Yo intermittent recovery level 1 test, a well-established and ecologically valid test widely used to mimic the high-intensity running bouts of soccer match-play. However, while these findings suggest that nitrate may be an effective ergogenic aid for team-sport players when consumed daily, it is currently unclear if the improvement in team-sport specific intermittent exercise performance can be achieved following a single bolus of dietary nitrate. Given the increasing interest and use of dietary nitrate as an ergogenic aid by team-sport players, establishing the shortest period of supplementation required to elicit an ergogenic effect is important in order to guide athletes on optimal supplementation strategies.

Given that a single bolus of dietary nitrate has previously been shown to improve exercise tolerance and endurance exercise performance, and an improved Yo-Yo IR1 performance has been observed after chronic nitrate supplementation, the investigator hypothesizes that acute (2 h) and short-term (4 days) nitrate supplementation will significantly elevate nitric oxide activity (measured as an increase in plasma nitrite concentration and skeletal muscle nitrate concentration) and improve performance during the Yo-Yo IR1 test (measured as an increased in distance covered (m) during the test at the point of volitional exhaustion) to a similar extent, when compared to a placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male, physically active, intermittent team sport players, in self-reported good general health as assessed by the standard procedures described below and specifically meeting the following: blood pressure (BP), systolic 100-135 mmHg and diastolic 60-90 mmHg, and; body mass index (BMI) 16-29.9.
2. 18-35 years of age
3. Participants must participate in an intermittent exercise based sport (e.g. soccer, rugby, hockey), at a competitive level (i.e. competes in officiated matches/games).
4. Understanding of the procedures to be undertaken as part of the study
5. Willingness to participate in exercise testing and follow supplementation guidelines and other instructions provided by the experimenter
6. Informed, voluntary, written consent to participate in the study

Exclusion Criteria:

1. Known pulmonary, cardiovascular or metabolic disease
2. Food allergies including phenylketonurea (PKU)
3. Current regular use of any dietary supplement (excluding macronutrient based supplements) or previous use of any dietary supplement in the past 6 months that is known to have a lasting effect.
4. Blood donation within 3 months prior to the start of the study
5. Substance abuse within 2 years of the start of the study
6. Smoking
7. Any prescription and non-prescription medication which may impact saliva production (antidepressants, diuretics, analgesics, antihistamines, anti-hyper/hypo-tensives, anti-anxiety, appetite suppressants).
8. Current or previous use of phosphodiesterase 5 (PDE5) inhibitors.
9. Participation in another clinical trial within past 4 weeks and/or participation in a PepsiCo trial within the last 6 months.
10. Chronic use (6 months) of any antibacterial mouthwash products.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Distance covered during high-intensity intermittent exercise performance | 4 days
Distance covered during high-intensity intermittent exercise performance | 2 hours

SECONDARY OUTCOMES:
Plasma nitrate concentrations | 4 days
Nitrite concentrations | 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University of Exeter, Sport and Health Sciences department,, Exeter, United Kingdom